CLINICAL TRIAL: NCT02836548
Title: HDAC Inhibitor Vorinostat in Resistant BRAF V600 Mutated Advanced Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16VOM
Record Dates: First submitted 2016-06-24; First posted 2016-07-19 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2018-10

CONDITIONS: Melanoma; Skin Neoplasms
Keywords: advanced melanoma; BRAF V600 mutation; vorinostat; HDAC inhibitor
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Vorinostat; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vorinostat (Experimental): Vorinostat 360 mg once daily
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — vorinostat 360 milligram once daily
  Other Names: HDAC inhibitor

SUMMARY:
This is a mono-center open-label proof-of-concept pharmacologic study to explore the efficacy and safety of vorinostat in advanced BRAF mutated melanoma, which became resistant for BRAF-inhibitors or the combination of BRAF- and MEK-inhibitors.

DETAILED DESCRIPTION:
Activating mutations in the BRAF gene are present in about 50% of human melanomas. BRAF inhibitors (BRAFi) inhibit the serine-threonine protein kinase BRAF, which plays a dominant role in the MAPK pathway influencing cell growth. MEK inhibitors (MEKi) inhibit MEK1 and MEK2, two regulatory proteins downstream of BRAF.

The clinical benefit of this treatment is limited due to development of drug resistance in 6-8 months for treatment with BRAFi and 9-14 months for treatment with BRAFi in combination with MEKi.This is often associated with secondary mutations in the MAPK pathway leading to re-activation of the pathway.Withholding from treatment with BRAFi and/or MEKi leads to a reversible hyperactivation of the MAPK pathway, causing a transient growth arrest. Chronic proliferation and growth arrest occur when there is a persistent hyperactivation of the MAPK pathway. Treatment of BRAFi and/or MEKi resistant melanoma with vorinostat, a histone deacetylase inhibitor (HDACi), leads to persistent hyperactivation of the pathway and a state of growth arrest with hallmarks of oncogene induced senescence.In these studies in mice with BRAFi resistant BRAF V600 mutated melanoma switch from a BRAFi to the HDACi vorinostat resulted in complete disappearance of the tumor after two months of treatment.

HDACi cause accumulation of Reactive Oxygen Species (ROS) leading to apoptosis and upregulation of the MAPK-pathway. As seen by Wang et al hyperactivation of the MAPK-pathway is an important milestone in the anti-tumor treatment of BRAF V600 melanoma.

This is a phase I, single-center, single-arm, non-randomized, open-label, clinical pharmacological proof of principal study to determine the safety of vorinostat as anti-tumor therapy in patients with advanced resistant BRAF V600 mutated melanoma. A total of 21 evaluable patients with BRAF V600 mutated melanoma who developed resistance to BRAFi and/or BRAFi+MEKi after at least 4 weeks of PR or CR response will be enrolled in this study. Vorinostat will be given at a single daily dose of 360 mg derived from the established and registered dose for treatment of cutaneous T-cell lymphoma. Treatment will be continuous in cycles of 28 days and doses will be reduced in steps of 90 mg per dose-reduction in case of unacceptable safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of advanced melanoma with BRAF V600 mutation;
2. Progression of disease, according to RECIST 1.1, while on treatment with BRAFi, such as vemurafenib or dabrafenib; or a combination of BRAF - and MEK inhibitors, such as trametinib and dabrafenib;
3. Previous documented response (partial or complete) for at least 4 weeks to treatment with BRAFi and/or BRAFi+MEKi;
4. Start with vorinostat treatment within a maximum period of 1 week after discontinuation of BRAFi and/or BRAFi+MEKi.

   The BRAFi and/or BRAFi+MEKi can be continued after progression to provide sufficient time to perform baseline assessments;
5. Age ≥ 18 years;
6. Able and willing to give written informed consent;
7. WHO performance status of 0, 1 or 2;
8. Able and willing to undergo blood sampling for PK and PD analysis;
9. Life expectancy ≥ 3 months allowing adequate follow up of toxicity evaluation and antitumor activity;
10. Evaluable disease according to RECIST 1.1;
11. Minimal acceptable safety laboratory values

    * ANC of ≥ 1.5 x 109 /L
    * Platelet count of ≥ 100 x 109 /L
    * Hemoglobin ≥ 6.0 mmol/L
    * Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALAT and ASAT ≤ 2.5 x ULN, or in case of liver metastases ALAT and ASAT ≤ 5 x ULN
    * Renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula, or MDRD).
12. Negative pregnancy test (urine/serum) within 72 hours before receiving the first dose of study medication for female patients with childbearing potential;
13. Able and willing to undergo fresh histological tumor sampling prior to start, upon treatment and upon progression of vorinostat.

Exclusion Criteria:

1. Any treatment with investigational drugs, except BRAFi and MEKi, within 28 days prior to receiving the first dose of investigational treatment; or 21 days for standard chemotherapy and immunotherapy;
2. Patients who have had previous treatment with vorinostat or other HDAC inhibitors;
3. Leptomeningeal disease;
4. Symptomatic brain metastasis. Patients previously treated or untreated for the condition and/or who are asymptomatic in the absence of corticosteroid therapy are allowed to enroll. Patients are not permitted to receive enzyme inducing anti-epileptic drugs or corticosteroids;
5. Clinical progression of melanoma in the first week of discontinuation of BRAFi or BRAFi/MEKi;
6. Woman who are pregnant or breast feeding;
7. Unreliable contraceptive methods. Both men and women enrolled in this trial must agree to use a reliable contraceptive method from screening until 30 days after the last dose of study medication (adequate contraceptive methods are: oral or injected or implanted hormonal methods of contraception, condom, sterilization, other barrier contraceptive measures preferably in combination with condoms, true abstinence);
8. Radiotherapy within the last 4 weeks prior to receiving the first dose of investigational treatment; except 1x8 Gray for pain palliation;
9. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
10. Patients with a known history of hepatitis B or C;
11. Recent myocardial infarction (< 6 months before receiving the first dose of study medication) or unstable angina;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-06; Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Anti-tumor response rate in at least 30% of the treated patients. | CT scan every 6 weeks up to 24 months and monthly phone call until start of subsequent anticancer therapy or until all patients have been followed up for at least 24 months or have been lost to follow up, whichever occurs first.
  Overall response rate measured by RECIST v 1.1.

SECONDARY OUTCOMES:
Tolerability (incidence and severity of adverse events per CTCAE v4.03) | Up to 28 days after last drug intake
  Incidence and severity of adverse events per CTCAE v4.03
progression free survival (PFS) per RECIST v1.1 | CT scan every 6 weeks up to 24 months and monthly phone call until start of subsequent anticancer therapy or until all patients have been followed up for at least 24 months or have been lost to follow up, whichever occurs first
  PFS measured by RECIST v 1.1.
Overall survival (ORR) per RECIST v1.1 | CT scan every 6 weeks up to 24 months and monthly phone call until start of subsequent anticancer therapy or until all patients have been followed up for at least 24 months or have been lost to follow up, whichever occurs first
  ORR measured by RECIST v 1.1.
Plasma concentrations of vorinostat | On day 1 and 15 in cycle 1(each cycle is 28 days).
  Plasma concentrations of vorinostat will be measured at day 1 and 15 in cycle 1 to determine pharmacokinetics and interindividual differences after a single dose and after multiple doses.
Determinants and mode of response -Target proteins | At baseline, cycle 1(each cycle is 28 days) day 1, day 15 and at treatment discontinuation (expected 6-9 months after start)
  Change in expression and/or phosphorylation status target proteins (e.g. pMEK, pERK, acetylated Histone 3) before, during and after treatment
Pharmacogenetics profiling to assess predictors of response and resistance- inducing mutations | before treatment, every 6 weeks up to 24 months and at treatment discontinuation (expected 6-9 months after start)
  Pharmacogenetic profiling to assess predictors of response and resistance-inducing mutations.

CONTACTS AND LOCATIONS:
Overall Officials: S Wilgenhof, MD, PhD, Principal Investigator — AVL-NKI
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huijberts S, Wang L, de Oliveira RL, Rosing H, Nuijen B, Beijnen J, Bernards R, Schellens J, Wilgenhof S. Vorinostat in patients with resistant BRAFV600E mutated advanced melanoma: a proof of concept study. Future Oncol. 2020 Apr;16(11):619-629. doi: 10.2217/fon-2020-0023. Epub 2020 Mar 3. PMID 32125175